CLINICAL TRIAL: NCT00226694
Title: Alcohol and Gender Effects on Stress Circuit Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: NIAAAANH013307; R01AA013307 (NIH); NIH R01 AA013307-01
Record Dates: First submitted 2005-09-23; First posted 2005-09-27 (Estimated); Last update posted 2014-01-07 (Estimated); Status verified 2014-01

CONDITIONS: Alcoholism; Stress; Alcohol Dependence
Keywords: Alcoholism; Stress; Gender Differences; Addiction; Alcohol Dependence
MeSH Terms: conditions — Alcoholism; Behavior, Addictive | interventions — Citalopram; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Citalopram Group (Active Comparator): Subjects receive provocative tests with citalopram, dexamethasone/corticotropin-releasing hormone and placebo on 3 separate, counterbalanced occasions at monthly intervals.
  Interventions: Drug: Citalopram
- Placebo Group (Placebo Comparator): Subjects receive provocative tests with citalopram, dexamethasone/corticotropin-releasing hormone and placebo on 3 separate, counterbalanced occasions at monthly intervals.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Citalopram — Subjects receive provocative tests with citalopram, dexamethasone/corticotropin-releasing hormone and placebo on 3 separate, counterbalanced occasions at monthly intervals.
  Other Names: Celexa
  Arms: Citalopram Group
Other: Placebo — Subjects receive provocative tests with citalopram, dexamethasone/corticotropin-releasing hormone and placebo on 3 separate, counterbalanced occasions at monthly intervals.
  Other Names: Sugar Pill
  Arms: Placebo Group

SUMMARY:
The purpose of this study is to look at the stress hormone response to medication-induced stress and a placebo (an inactive compound) in non-drinking, recovering male and female alcoholics, with a specific emphasis on the differences between men and women in the two recovering alcoholic groups.

DETAILED DESCRIPTION:
Women and men differ in the ways stress affects the development and maintenance of alcoholism. However, no published studies in alcohol dependent patients have examined sex differences in stress responsiveness that most likely mediate these effects and influence the clinical course and treatment of the disorder.

The long-range goal of this research program is to define aspects of the neural, genetic and environmental mechanisms differentially regulating the stress response in alcohol dependent women and men. The proposed study extends prior work revealing sex-dependent alterations in basal and serotonin-induced stress hormone concentrations in abstinent alcoholics. Our central hypothesis is that sex differences in serotonin function or HPA sensitivity conspire with genetically influenced alterations in serotonin signaling to produce maladaptive stress responses in some alcoholic women. These altered stress responses may serve as the target of novel, sex-specific pharmacotherapies.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written consent.
* Are actively engaged in a recovery program for alcoholism;
* Have a current (within the past 12 months) diagnosis of DSM-IV alcohol dependence in early- (modified to a minimum of 4 months) full remission; and
* Are residing in a controlled sober living environment; and
* Agree to provide at least one collateral informant who knows the subject well and can attest to their sobriety (recovering alcoholics only).

Exclusion Criteria:

* Have evidence of any clinically significant laboratory evidence of hematologic, hepatic, cardiovascular, renal, pulmonary, thyroid or other endocrine disease;
* Are taking oral contraceptives or other hormonal replacements (e.g., estrogen or progesterone);
* Are pregnant, or planning to become pregnant during the next 9 months;
* Have taken other psychotropic drugs (including SSRIs, MAO inhibitors and other antidepressants, antipsychotics, mood stabilizers, non-benzodiazepine anxiolytics or hypnotics) within 6 weeks of the first laboratory session;
* Have taken any investigational drug within 90 days of the first laboratory session; or
* Are making efforts to quit smoking or have taken any pharmacotherapies for smoking cessation (i.e., bupropion, nicotine-replacement patches or gum; clonidine, buspirone) within 90 days of the first laboratory session.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2003-09; Primary Completion 2011-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
stress | month

CONTACTS AND LOCATIONS:
Overall Officials: Robert M. Anthenelli, MD, Principal Investigator — US Department of Veterans Affairs
Locations (1):
- The Department of Veterans Affairs / Veterans Healthcare System of Ohio, Cincinnati, Ohio, United States